CLINICAL TRIAL: NCT02004470
Title: Lavage and Suction of the Right Upper Quadrant to Reduce Post Laparoscopic Shoulder Pain: A Randomized Controlled Trial
Brief Title: Lavage and Suction of the Right Upper Quadrant to Reduce Post Laparoscopic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LAS-37405
Record Dates: First submitted 2013-11-15; First posted 2013-12-09 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Shoulder Pain
Keywords: post laparoscopic shoulder pain; active suction; lavage and suction; right shoulder pain; post operative shoulder pain
MeSH Terms: conditions — Shoulder Pain | interventions — Suction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Passive exsufflation (No Intervention): Will not actively suction carbon dioxide from abdomen. Open laparoscopic trocars and allow C02 to passively empty from abdomen.
- Active lavage and suction (Experimental): This step is already employed in many ongoing surgeries where normal saline will be used to lavage the right upper quadrant and then will be suctioned out to remove as much Carbon dioxide from the patient's abdomen and to therefore decrease postoperative pain.
  Interventions: Procedure: Active lavage and suction

INTERVENTIONS:
Procedure: Active lavage and suction — Active lavage and suction of the right upper quadrant will be performed as the laparoscopic procedure is about to be terminated.
  Arms: Active lavage and suction

SUMMARY:
The use of laparoscopy in gynecologic surgery has been well established to decrease morbidity, blood loss, hospital stay, and post-operative pain when compared to traditional open abdominal surgery. However, the laparoscopic technique is associated with post-operative shoulder pain.

We hypothesize that a combination of intraperitoneal saline lavage and active suction removal of carbon dioxide gas from the right upper quadrant of the abdomen will decrease incidence of post-laparoscopic shoulder pain when compared to passive exsufflation of carbon dioxide gas.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patient
* Female
* Age 18-75
* must undergo laparoscopic surgery
* willing to participate in the study

Exclusion Criteria:

* Male patients
* Under 18 or older than 75
* Laparoscopic procedures that get converted to laparotomy
* Intraoperative hemorrhage more than 500 cc
* Patients with active joint disease
* History of shoulder surgery
* Intraoperative laceration to the liver
* Malignancy
* Long term daily narcotic use
* Chronic right upper quadrant/ shoulder pain
* Pregnancy
* History of dementia, Alzheimers, stroke or other condition causing altered mental status

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 12 hours
  We will assess pain scores based on visual analog score from 1-10 at 12 hours postoperatively.
Pain Score | 24 hours
  We will assess a pain score at 24 hours post operatively based on a visual analog score of 1-10
Pain Score | 48 hours
  We will assess a pain score based on a visual analog score of 1-10 at 48 hours post operatively.

SECONDARY OUTCOMES:
operative time | 24 hours
  We will assess how long each surgery takes to complete.
blood loss | 6 hours
  We will assess intraoperative blood loss.
analgesic use | 7 days
  We will assess total analgesic, iv and oral used over the course of 7 days postoperatively.
Anti emetic use | 48 hours
  Total amount of intravenous and oral narcotic used postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Hadiashar, MD, Principal Investigator — University of Tennessee Chattanooga College of Medicine
Locations (4):
- United States (4):
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Parkridge East Hospital, Chattanooga, Tennessee
  - Erlanger East Hospital, Chattanooga, Tennessee

REFERENCES:
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Result] Tsai HW, Wang PH, Yen MS, Chao KC, Hsu TF, Chen YJ. Prevention of postlaparoscopic shoulder and upper abdominal pain: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):526-531. doi: 10.1097/AOG.0b013e318283fcca. PMID 23635614
- [Result] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749